CLINICAL TRIAL: NCT05128903
Title: Quantitative Assessment of Radiation-induced Neuroinflammation - A Proof of Principle Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QARIN1
Record Dates: First submitted 2021-11-05; First posted 2021-11-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Brain Tumor; Medulloblastoma
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants who meet the eligibility criteria in the study will receive Translocation Protein (TSPO) Positron Emission Tomography (PET) for longitudinal, quantitative assessment of brain neuroinflammation following whole brain radiation therapy.
  Interventions: Drug: [18F]DPA714

INTERVENTIONS:
Drug: [18F]DPA714 — Intravenous injection
  * Before or within 2 weeks of starting radiation therapy
  * Before starting chemotherapy
  * 1 year after the start of radiation therapy Timing cont.
  * 1.5 to 2 years after the start of radiation therapy

SUMMARY:
QARIN 1 is a study of [18F]DPA-714 Translocation Protein (TSPO) Positron Emission Tomography (PET) for longitudinal, quantitative assessment of brain neuroinflammation following whole brain radiation therapy. This TSPO PET, uses a radioactive tracer. An optional MRI (magnetic resonance imaging) will also be performed to monitor brain microstructure damages induced by neuroinflammation.

Primary Objectives

* Assessment of temporal and regional variability of uptake of translocator protein (TSPO) positron emission tomography (PET) tracer.
* Regional variability will be assessed in medial temporal lobe, frontal lobe, and in white matter
* Temporal variability will be assessed by scanning each subject four-times: at baseline (before or within 2 weeks of start of radiation therapy), before start of chemotherapy, at 1 year from the initiation of the radiation therapy, and at 1.5-2 years from the initiation of the radiation therapy
* Correlation of radiation dose in specific brain regions with radiation induced neuroinflammation as measured by uptake of TSPO PET tracer.

Exploratory Objectives

* Assessment of radiation-induced brain microstructure injuries (RIBMI) in specific brain regions (medial temporal lobe, frontal lobe, and in white matter) using advanced magnetic resonance imaging (MRI) techniques.
* Association of radiation dose with MRI measures of RIBMI in these specific brain regions.
* Association of PET measures of RIN with MRI measures of RIBMI.
* Association of PET measure of RIN and MRI measures of RIBMI in specific regions of interest (ROI) with specific domain of neuro-cognition. For example, to investigate whether PET measure of RIN and MRI measures of RIBMI in hippocampal ROI have strongest association with episodic memory; whether frontal lobe cortical ROI are associated with attention and executive function.
* Association of a novel MRI based technique for assessment of RIN with TSPO PET.
* Association of the PET and MRI measure of neuroinflammation within 2- years of completion of radiation with delayed cognitive outcome that will be measured at 3, 4 and 5 years from the completion of radiation

DETAILED DESCRIPTION:
The participant will have 4 PET scans using a novel PET tracer that will help the investigators to quantify when and where in brain neuroinflammation happens following radiation therapy. The participant will receive the first PET scan either before your first dose of radiation therapy or within 2 weeks of the start of radiation therapy. The second PET scan will be obtained before starting chemotherapy. The third scan will be after 1 year of treatment.The final scan will be 1 and a half to 2 years after the start of treatment.The scan process will begin an hour or so after the participant has been given tracer by injection. The entire PET scan process lasts about 2 hours.

ELIGIBILITY:
Inclusion Criteria

* Participant is at least 8 years of age
* Participants with histologically confirmed medulloblastoma and are scheduled to receive 36 Gy craniospinal irradiation
* Participant and/or guardian can understand and is willing to sign a written informed consent document according to institutional guidelines
* Subjects have either have high-affinity or mixed-affinity TSPO binding sites as determined by the single-nucleotide polymorphism (SNP) rs6971 in the TSPO gene.

Exclusion Criteria:

* Participants with a large pseudomeningocele (>4 cm in size) at the surgical site, complications from ventricular access (evidenced by hemorrhage and/or enhancement along the catheter), large subdural effusion in the supra-tentorial compartment (>1 cm in the maximum transverse dimension). All of these are expected to induce inflammation.
* Female participants of childbearing age must not be lactating due to theoretical potential harm to the infant from exposure to radiation.
* Subjects with low-affinity TSPO binding sites as determined by the single-nucleotide polymorphism (SNP) rs6971 in the TSPO gene.
* Pregnant subjects.
* Patients needing sedation for the PET scans or optional MRI scans.
* Participants with a diagnosis of recurrent medulloblastoma.

Ages: 8 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 22 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2035-10-26 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
SUVr | follow up 1: up to 13 weeks after radiation therapy
  SUVr values for dorsolateral prefrontal cortex comparing baseline vs. follow up 1
SUVr | follow up 1 : up to 13 weeks after radiation therapy
  SUVr values for medial prefrontal cortex comparing baseline vs. follow up 1
SUVr | follow up 1 : up to 13 weeks after radiation therapy
  SUVr values for hippocampus comparing baseline vs. follow up 1.
SUVr | follow up 1 : up to 13 weeks after radiation therapy
  SUVr values for Corpus callosum comparing baseline vs. follow up 1.
SUVr | follow up 1 : up to 13 weeks after radiation therapy
  SUVr values for corticospinal tract comparing baseline vs. follow up 1.
SUVr | follow up 1 : up to 13 weeks after radiation therapy
  SUVr values for superior longitudinal fasciculus comparing baseline vs. follow up 1
SUVr | follow up 2: up to 53 weeks after radiation therapy
  SUVr values for dorsolateral prefrontal cortex comparing baseline vs. follow up 2.
SUVr | follow up 2: up to 53 weeks after radiation therapy
  SUVr values for medial prefrontal cortex comparing baseline vs. follow up 2.
SUVr | follow up 2: up to 53 weeks after radiation therapy
  SUVr values for hippocampus comparing baseline vs. follow up 2.
SUVr | follow up 2: up to 53 weeks after radiation therapy
  SUVr values for Corpus callosum comparing baseline vs. follow up 2.
SUVr | follow up 2: up to 53 weeks after radiation therapy
  SUVr values for corticospinal tract comparing baseline vs. follow up 2.
SUVr | follow up 2: up to 53 weeks after radiation therapy
  SUVr values for superior longitudinal fasciculus comparing baseline vs. follow up 2.
SUVr | follow up 3: up to 2 years after radiation therapy
  SUVr values for dorsolateral prefrontal cortex comparing baseline vs. follow up 3.
SUVr | follow up 3: up to 2 years after radiation therapy
  SUVr values for medial prefrontal cortex comparing baseline vs. follow up 3.
SUVr | follow up 3: up to 2 years after radiation therapy
  SUVr values for hippocampus comparing baseline vs. follow up 3.
SUVr | follow up 3: up to 2 years after radiation therapy
  SUVr values for Corpus callosum comparing baseline vs. follow up 3
SUVr | follow up 3: up to 2 years after radiation therapy
  SUVr values for corticospinal tract comparing baseline vs. follow up 3.
SUVr | follow up 3: up to 2 years after radiation therapy
  SUVr values for superior longitudinal fasciculus comparing baseline vs. follow up 3.

CONTACTS AND LOCATIONS:
Overall Officials: Asim Bag, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St.Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols